## Early Feasibility Prospective Open-Label Study to Assess the Function of a Novel Pessary for the Non-Surgical Management of Pelvic Organ Prolapse

| <b>Protocol Number:</b> | CP-001 |
|---|---|
| NCT Number: | NCT04275089 |
| Sponsor: | Reia, LLC ("Reia") |
| | 331 River Road |
| | Lyme, NH 03768 |
| Medical Monitor: | Paul Hanissian, MD |
| | 331 River Road |
| | Lyme, NH 03768 |
| <b>Principle Investigator:</b> | Kris Strohbehn, MD |
| Study Site: | Department of Obstetrics and Gynecology |
| | Dartmouth-Hitchcock Medical Center |
| | One Medical Center Drive |
| | Lebanon, NH 03756 |
| | Kris.Strohbehn@Hitchcock.org |
| | Direct phone number for office of the PI: 603 653-9312 |
| | 24-hour phone number: 603 650-5000 |
| <b>Document Date:</b> | 2/17/2020 |

## **Statistical Design and Power**

Recognizing that formal statistical procedures and power analyses are not the main focus of an early feasibility trial for a medical device, a few points will be made about the choice of 15 subjects. As reported by Cundiff et al. (2007), of 57 women initially successfully fitted with the Gellhorn pessary, within a week 21 had to be refitted which is a short-term fitting failure rate of about 37%. A 95% confidence interval about this proportion using an exact binomial test ranges from 24% to 51%. We can record the number of short-term failures in our preliminary study and compare our rate to Cundiff et al. If 4 of 15 (27%) of our subjects or fewer have to be refit, we could reject the null hypothesis of a short-term failure rate of .51 or greater at p < .05. Or, from a power perspective, if our true short-term failure rate was 21% or lower, power would be .81 or higher to reject the null hypothesis that our true failure rate is 51% or greater. This would give us another perspective on how fitting our new pessary compares to fitting existing pessaries.